CLINICAL TRIAL: NCT06746480
Title: A Single-Arm, Multicenter, Open-Label Phase IIa Clinical Study to Evaluate the Efficacy and Safety of VG161 in the Treatment of Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Clinical Study of VG161 in Advanced Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CNBG-Virogin Biotech (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG161-C201
Record Dates: First submitted 2023-02-19; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Advanced Intrahepatic Cholangiocarcinoma
Keywords: Advanced intrahepatic cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): 1.0 × 10^8 PFU/day per cycle, intratumoral injection for 3 consecutive days in 28-day cycles.
  Interventions: Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell))

INTERVENTIONS:
Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)) — Intratumoral injection only. The dosing date is Days 1 through 3.
  Other Names: VG161

SUMMARY:
VG161 is a recombinant human-IL12/15/PDL1B oncolytic HSV-1 Injectable. This trial is a single-agent, single-arm, multicenter, open-label design clinical trial for advanced intrahepatic cholangiocarcinoma who have failed standard therapy. To evaluate the efficacy of VG161 administered by ultrasound or CT-guided intratumoral injection in patients with advanced intrahepatic cholangiocarcinoma, with the primary outcome measure being objective response rate (ORR).

DETAILED DESCRIPTION:
The trial was conducted in two phases, and in the first phase, a total of 20 subjects were enrolled (per efficacy assessment analysis set). If 5 or more of the 20 subjects in Stage I achieve an objective response, i.e., the overall ORR is greater than 4/20, it suggests that the drug warrants further investigation and no additional subjects are required to enter Stage II. If only 1 or no subject out of 20 had an objective response, the trial was stopped, indicating that the trial drug had no apparent effect. Otherwise, continue to enter Stage II, add 13 subjects (as per efficacy evaluation analysis set), and the total number of subjects reaches 33. If 5 or more of 33 subjects achieve objective response, i.e., the overall ORR is greater than 4/33, it indicates that the drug has good anti-tumor efficacy and is worthy of entering confirmatory clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must fully understand and give informed consent to this study before the trial, and voluntarily sign a written informed consent form.

  2. aged 18 to 75 years (inclusive), male or female. 3. patients with histologically or cytologically confirmed advanced intrahepatic cholangiocarcinoma.

  4. According to the Guidelines for the Diagnosis and Treatment of Biliary Malignant Tumors (CSCO), patients must have previously received at least systemic first-line therapy for advanced intrahepatic cholangiocarcinoma and failed, or cannot tolerate treatment. Patients who received preoperative neoadjuvant chemotherapy or postoperative adjuvant chemotherapy were counted as having failed first-line treatment if disease progression occurred during chemotherapy or within 6 months after stopping chemotherapy; 5. According to RECIST 1.1 criteria, one or more CT examinations are determined to be measurable and meet the requirements for the volume administered for the first injection, tumor lesions and/or metastases (the injected lesions should preferably be the main tumor burden lesions) that can be injected under ultrasound or CT guidance, and the baseline longest diameter of the injected lesions (lymph node lesions are short diameters) is > 1.5 cm.

  6. Herpes simplex virus type I (HSV-1) antibody test results (HSV-1 IgG or HSV-1 IgM) are positive.

  7. ECOG performance score 0-1. 8. Expected survival time of more than 3 months. 9.Adequate organ function:
  1. Blood routine (no blood transfusion or colony-stimulating factor treatment within 14 days): ANC ≥ 1.5 × 109/L, PLT ≥ 75 × 109/L, Hb ≥ 85 g/L;
  2. Liver function: TBIL ≤ 1.5 × ULN, ALT ≤ 3 × ULN, AST ≤ 3 × ULN;
  3. Child-Pugh A-B;
  4. Renal function: Cr ≤ 1.5 × ULN, and creatinine clearance ≥ 45ml/min (calculated according to Cockcroft-Gault formula);
  5. Coagulation function: activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN, international normalized ratio (INR) ≤ 1.5 × ULN; 10.Eligible patients of childbearing potential (men and women) must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) during the trial and for at least 90 days after the last dose; female patients of childbearing potential must have a negative blood pregnancy test within 7 days prior to enrollment.

     Exclusion Criteria:
* 1. received chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor drugs within 4 weeks before the first use of the study drug, of which oral fluorouracil and small molecule targeted drugs were within 2 weeks before the first use of the study drug or within 5 half-lives of the drug (whichever was longer).

  2. Patients who have received transcatheter arterial chemoembolization (TACE) within 4 weeks before the first use of the study drug.

  3. Received other clinical trial drugs that are not approved for marketing within 4 weeks before the first use of the study drug.

  4. Major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks before the first dose of study drug.

  5. Have received a vaccine within 4 weeks prior to the first dose of study drug.

  6. Patients who have received systemic corticosteroids (prednisone > 10 mg/day or equivalent doses of the same class of drugs) or other immunosuppressive agents within 14 days before the first dose of study drug; except for the following: topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term corticosteroids (≤ 10 mg prednisone equivalent) for prophylaxis (e.g., prevention of contrast agent allergy).

  7. The adverse reactions of previous anti-tumor treatment have not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except alopecia and other toxicities that are judged by the investigator to have no safety risk); 8. Patients with central nervous system metastasis, spinal cord metastasis and/or spinal cord compression.

  9. in the herpes simplex virus recurrence and infection period, and there are corresponding clinical manifestations, such as oral herpes labialis, herpetic keratitis, herpetic dermatitis, genital herpes and so on.

  10. other active uncontrolled infections. 11. History of immunodeficiency, including positive HIV antibody test and positive Treponema pallidum antibody test.

  12. Patients with active chronic hepatitis B or active hepatitis C. (Except hepatitis B virus carriers, hepatitis B virus stable after drug treatment [HBV-DNA negative or < 500 IU/ml] and cured hepatitis C patients [HCV RNA negative]) 13. History of serious cardiovascular disease:
  1. Ventricular arrhythmia requiring clinical intervention;
  2. QTc interval > 480 ms;
  3. Acute coronary syndrome, congestive heart failure, stroke or other Grade III and above cardiovascular events within 6 months before the first use of study drugs;
  4. New York Heart Association (NYHA) functional classification ≥ II or left ventricular ejection fraction (LVEF) < 40%;
  5. Uncontrolled hypertension after treatment (judged by the investigator); 14. Patients with active, or have had and have the possibility of relapse of autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.); except for clinically stable autoimmune thyroiditis, autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone, type I diabetes treated with stable doses of insulin, vitiligo or recovered childhood asthma/allergy, without any intervention in adults.

  15. Having received immunotherapy and have experienced immune-related adverse events (irAEs) such as immune-related pneumonia and myocarditis, which may affect the safety of the investigational drug as judged by the investigator.

  16. Known alcohol or drug dependence. 17. Patients with mental disorders or poor compliance. 18. Pregnant or lactating women. 19. The investigator believes that the subject has other serious systemic diseases or other reasons and is not suitable for this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-03-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 27 months
  Efficacy evaluation endpoint measures will be evaluated according to iRECIST criteria and refer to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
PFS | 27 months
  Evaluate medium Progression Free Survival by iRECIST
6-month survival rates (OS rate) | 33 months
  Evaluate Overall Survival rate
6-month overall survival (OS) | 33 months
  Overall Survival
12-month survival rates (OS rate) | 39 months
  Evaluate Overall Survival rate
12-month overall survival (OS) | 39 months
  Overall Survival
DOR | 27 months
  Evaluate Disease Control Rate by iRECIST
peripheral blood lymphocyte subsets (CD3 +, CD4 +, CD8 +, CD4 +/CD8 + ratio, NK, CD19 +, CD56 + cells) | 27 months
  Concentration of CD3+, CD4+, CD8+, CD4 +/CD8 + ratio, NK, CD19 +, CD56 + cells
cytokines (IL-6, TNF-α, IFN-γ) | 27 months
  Concentration of IL-6, TNF-α, IFN-γ
T cell-related parameters (PD-L1, PD-1, CD69, CD8 + Ki67high) | 27 months
  Concentration of PD-L1, PD-1, CD69, CD8 + Ki67high
Safety indicators：laboratory tests results | 27 months
  Incidence of abnormal laboratory tests results

OTHER OUTCOMES:
Exploratory Endpoints | 27 months
  Single-cell sequencing was performed on tumor biopsy samples to explore biomarkers predictive of clinical response to VG161.

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No